CLINICAL TRIAL: NCT02401334
Title: Feasibility Study of the Antimicrobial Hernia Repair Device for Repair of Ventral or Incisional Hernia
Brief Title: Antimicrobial Hernia Repair Device Clinical Study
Acronym: AMEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-10
Record Dates: First submitted 2015-03-24; First posted 2015-03-27 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Ventral Hernia; Incisional Hernia
MeSH Terms: conditions — Hernia, Ventral; Incisional Hernia

ARMS (1):
- Hernia Repair (Experimental): Surgical repair for hernia with implantation of the Cook® Antimicrobial Hernia Repair Device.
  Interventions: Device: Cook® Antimicrobial Hernia Repair Device

INTERVENTIONS:
Device: Cook® Antimicrobial Hernia Repair Device — Device containing an antimicrobial to reinforce soft tissue during ventral or incisional hernia repair in clean-contaminated, contaminated, and dirty-infected

SUMMARY:
This prospective clinical study will evaluate the safety and efficacy of the Cook® Antimicrobial Hernia Repair Device containing an antimicrobial to reinforce soft tissue during ventral or incisional hernia repair in clean-contaminated, contaminated, and dirty-infected (i.e., Class II, Class III, and Class IV) surgical fields. Up to 30 patients will be treated with the Cook® Antimicrobial Hernia Repair Device and patients will be followed for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient presents with a ventral or incisional hernia that is to be surgically corrected using open repair technique

Exclusion Criteria:

* Body Mass Index (BMI) < 25.
* Body weight < 45 kg
* Glycosylated Hemoglobin (Hgb A1c) > 10%
* Albumin < 2.5 g/dL or pre-albumin < 5.0 mg/dL
* Renal insufficiency, as determined by an estimated glomerular filtration rate (GFR) < 60 mL/min/1.73 m2
* Known allergies to study device components
* Other relevant exclusion criteria apply

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-06; Primary Completion 2018-01-25 (Actual); Study Completion 2018-01-25 (Actual)

PRIMARY OUTCOMES:
Incidence of Surgical Site Infection | 6 months

SECONDARY OUTCOMES:
Incidence of procedural or post-operative adverse events related to the study device or procedure (i.e., Permanence of hernia repair, as determined by hernia recurrence). | 12 months

CONTACTS AND LOCATIONS:
Locations (4):
- Canada (2):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
- United Kingdom (2):
  - Salford Royal Hospital, Salford, England
  - Royal Liverpool Hospital, Liverpool

REFERENCES:
- [Derived] Minor S, Brown CJ, Rooney PS, Hodde JP, Julien L, Scott TM, Karimuddin AA, Raval MJ, Phang PT. Single-stage repair of contaminated hernias using a novel antibiotic-impregnated biologic porcine submucosa tissue matrix. BMC Surg. 2020 Mar 30;20(1):58. doi: 10.1186/s12893-020-00715-w. PMID 32228664